CLINICAL TRIAL: NCT06466616
Title: Efficacy of Applying Shock Waves Combined With Leg Stretching in Patients With Plantar Fasciitis: A Randomized Controlled Trial
Brief Title: Shock Waves Therapy Combined With Leg Stretching in Patients With Plantar Fasciitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Guillem Serrabassa Ureña, Principal investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IDCES-08969382A
Record Dates: First submitted 2024-06-10; First posted 2024-06-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Plantar Fascitis
Keywords: shockwave therapy; stretching; pain; disability; activity limitation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Stretching (Experimental): This group is going to realize 3 sessions of ESWT plus an 8 weeks stretching program.
  Interventions: Other: Real stretching
- Placebo Stretching (Placebo Comparator): This group is going to realize 3 sessions of ESWT plus an 8 weeks placebo stretching program.
  Interventions: Other: Placebo stretching

INTERVENTIONS:
Other: Real stretching — Aplying 3 sesions of ESWT in patients with plantar fasciitis in the zone of pain. Futhermore they are going to do a program of 8 weeks stretching of plantar fascia, gastrocnemius and hamstring muscle.
  Other Names: Extracorporeal Shock Wave Threatment
  Arms: Real Stretching
Other: Placebo stretching — Aplying 3 sesions of ESWT in patients with plantar fasciitis in the zone of pain. Futhermore they are going to do a program of 8 weeks placebo stretching of plantar fascia, gastrocnemius and hamstring muscle.
  Other Names: Extrecorporeal Shock Wave Threatment
  Arms: Placebo Stretching

SUMMARY:
The aim of this study is to evaluate the efficacy of a combination treatment consisting of ESWT and stretching of different muscles in the lower body compared to ESWT treatment alone in patients with plantar fasciitis.

DETAILED DESCRIPTION:
Background: Plantar fasciitis is the most common cause of pain in the heel of the foot, manifested by the presence of pain in the antero-internal part of the calcaneus. Currently, there is ample evidence of the efficacy of both shock waves and stretching in their treatment, however, no study has proven what results are obtained by combining the application of shock waves with stretching in different leg muscles.

Objectives: The main objective of the study is to compare the effects of OC treatment in conjunction with leg-length stretches against shock waves alone in reducing pain in patients with PF. The secondary objectives will be to observe the effects of both treatments on disability and activity limitation in both the short and medium term.

Materials and Methods: A double-blind randomized clinical trial will be conducted. A total of 52 subjects (26 in each group) will participate in the study, divided into one group that will undergo shockwave therapy plus real stretching (experimental group) and another that will undergo shockwave therapy plus placebo stretching (control group). The primary variable of the study will be pain, and secondary variables will include changes in disability and activity limitation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of pain in the medial area of the sole of the foot lasting 3 or more months.
* Being diagnosed with plantar fasciitis by one of the physical therapists participating in the study.
* Have a pain level equal to or greater than 3 on the Visual Analogue Scale (VAS).

Exclusion Criteria:

* Presence of bilateral plantar fasciitis.
* Signs of neurological abnormalities.
* Infections and malignant tumors.
* History of presence of dysfunction in the lower extremity.
* Pregnant women
* Have been treated with shock waves in the previous 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain intenisty VAS | Baseline (week 0), 8 weeks after baseline, 3 months after intervention and 12 months after intervention
  To evaluate the difference in pain after the intervention. We are going to use the Visual Analogue Scale, being 0 the better result and 10 the worst possible.
Pain intensity PSFP | Baseline (week 0), 8 weeks after baseline, 3 months after intervention and 12 months after intervention
  We are also to use the Pain Scale for Plantar Fasciitis in their section for pain measure. The minimum score is 0 (better) and the maximum 100 (worst).

SECONDARY OUTCOMES:
Disability | Baseline (week 0), 8 weeks after baseline, 3 months after intervention and 12 months after intervention
  To evaluate the difference in disability after the intervention. The Foot Function Index is going to be used to evaluate the disability, in its section intended for this. This scale gives a result in percent, the highest the percent is the worst.

OTHER OUTCOMES:
Activity limitation FFI | Baseline (week 0), 8 weeks after baseline, 3 months after intervention and 12 months after intervention
  To evaluate the difference in activity limitation after the intervention. The Foot Function Index is going to be used in order to evaluate the activity limitation, in its section intended for this. This scale gives a result in percent, the highest the percent is, the worst.
Activity limitation FAAM | Baseline (week 0), 8 weeks after baseline, 3 months after intervention and 12 months after intervention
  The Foot and Ankle Ability Measures is going to be used to evaluate activity limitation. It's section destinated to evaluate this item fives a number that goes from 0 to 84. This number must be divided by 100 to get de final percent. The highest the percent is, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Serrabassa Ureña, MSc, Principal Investigator — University of Alcalá; Tomás Gallego Izquierdo, PhD, Principal Investigator — University of Alcalá
Locations (1):
- University of Alcalá, Faculty of Nursing and Physiotherapy, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang YC, Chen SJ, Huang PJ, Huang HT, Cheng YM, Shih CL. Efficacy of Different Energy Levels Used in Focused and Radial Extracorporeal Shockwave Therapy in the Treatment of Plantar Fasciitis: A Meta-Analysis of Randomized Placebo-Controlled Trials. J Clin Med. 2019 Sep 19;8(9):1497. doi: 10.3390/jcm8091497. PMID 31546912
- [Background] Rhim HC, Kwon J, Park J, Borg-Stein J, Tenforde AS. A Systematic Review of Systematic Reviews on the Epidemiology, Evaluation, and Treatment of Plantar Fasciitis. Life (Basel). 2021 Nov 24;11(12):1287. doi: 10.3390/life11121287. PMID 34947818
- [Background] Sweeting D, Parish B, Hooper L, Chester R. The effectiveness of manual stretching in the treatment of plantar heel pain: a systematic review. J Foot Ankle Res. 2011 Jun 25;4:19. doi: 10.1186/1757-1146-4-19. PMID 21703003
- [Background] Rompe JD, Furia J, Cacchio A, Schmitz C, Maffulli N. Radial shock wave treatment alone is less efficient than radial shock wave treatment combined with tissue-specific plantar fascia-stretching in patients with chronic plantar heel pain. Int J Surg. 2015 Dec;24(Pt B):135-42. doi: 10.1016/j.ijsu.2015.04.082. Epub 2015 May 1. PMID 25940060
- [Background] Boonchum H, Bovonsunthonchai S, Sinsurin K, Kunanusornchai W. Effect of a home-based stretching exercise on multi-segmental foot motion and clinical outcomes in patients with plantar fasciitis. J Musculoskelet Neuronal Interact. 2020 Sep 1;20(3):411-420. PMID 32877978